CLINICAL TRIAL: NCT02670850
Title: A Model of Family Caregiving and Model-based Intervention Program for Family Caregivers of Patients With Mild Cognitive Impairment
Brief Title: Intervention Program for Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yea-Ing Lotus Shyu, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSC102-2314-B-182-051-MY3
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Family caregiver; Intervention program; Elders
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients received only routine hospital care
- Intervention group (Experimental): Patients received regular hospital routine care and model-based intervention program
  Interventions: Other: Family Caregiver Intervention Program

INTERVENTIONS:
Other: Family Caregiver Intervention Program — Family Caregiver Intervention Program included three components: introduction of mild cognitive impairment, maintain and improve cognitive function, and health management.
  Arms: Intervention group

SUMMARY:
Mild Cognitive Impairment (MCI) is a syndrome defined as a cognitive decline that is more severe than can be explained by an individual's age and education. One study in the United States found that MCI caregivers have experienced distress in association with caregiver burden. The prevalence of MCI for people age 65 and older ranges from 3% to 19%. Understanding the process of family caregiving provides a knowledge base for the health professionals when developing effective interventions. However, little is known about the phenomenon of family caregiving to patients with MCI in Taiwan.

Therefore, the purpose of the proposed study is to develop a theoretical model and a model-based intervention program for family caregivers of patients with MCI in Taiwan, and pilot test it in a clinical trial.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is a syndrome defined as a cognitive decline that is more severe than can be explained by an individual's age and education. One study in the United States found that MCI caregivers have experienced distress in association with caregiver burden. The prevalence of MCI for people age 65 and older ranges from 3% to 19%. Understanding the process of family caregiving provides a knowledge base for the health professionals when developing effective interventions. However, little is known about the phenomenon of family caregiving to patients with MCI in Taiwan.

Therefore, the purpose of the proposed study is to develop a theoretical model and a model-based intervention program for family caregivers of patients with MCI in Taiwan, and pilot test it in a clinical trial.

To conduct a small scale pilot randomized control trial (total N = 60; 30 in each group) to pilot test the intervention program. The intervention group will receive the caregiver training program, and the control group received printed sheets with general information on MCI and dementia such as the causes, courses and symptoms. At 1 month, 3 months, and 6 months after the intervention group will complete the two-session training program, both groups will receive a follow-up assessment for preparedness, HRQoL and depressive symptoms. To minimize attrition, caregivers in both groups will receive monthly follow-up phone calls from the first to the sixth month. Changes in outcome variables will be analyzed using hierarchical linear models, in order to provide a reference for further formal clinical trial.

ELIGIBILITY:
Patients' Inclusion Criteria:

* Age 65 years or older
* Being diagnosed as having MCI by a neurologist or a psychiatris
* Being cared for in a home setting

Patients' Exclusion Criteria:

* Terminally ill

Caregivers' Inclusion Criteria:

* Age 20 years or older
* Assuming primary responsibility for the care of the frail elderly person

Caregivers' Exclusion Criteria:

* Terminally ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Caregivers' preparedness was measured by the 10-item Caregiver Preparedness Scale. | 6 months

SECONDARY OUTCOMES:
Caregivers' competence was measured by the 17-item Competence Scale. | 6 months
Caregivers' quality of life was measured by the The 36-Item Short Form Health Survey (SF-36). | 6 months
Caregivers' depressive symptoms was measured by the the Center for Epidemiologic Studies Depression Scale. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No